CLINICAL TRIAL: NCT06591572
Title: Efficacy and Safety Assessment of Single-port Robotic Transanal Total Mesorectal Excision for Mid and Low Rectal Cancer: a Phase 2a Trial Based on the IDEAL Framework
Brief Title: Single-port Robotic Transanal Total Mesorectal Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPORTS-01
Record Dates: First submitted 2024-08-11; First posted 2024-09-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer Patients
Keywords: Single-port robotic; transanal total mesorectal excision; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-port robotic transanal total mesorectal excision (Experimental): Single-port robotic transanal total mesorectal excision
  Interventions: Procedure: Single-port robotic transanal total mesorectal excision

INTERVENTIONS:
Procedure: Single-port robotic transanal total mesorectal excision — Rectal resection by transanal TME with single-port robotic surgery

SUMMARY:
This is a phase 2a clinical trial based on the IDEAL framework to evaluate the safety, feasibility and clinical efficacy of single-port robotic transanal total mesorectal excision (SPr-taTME )surgery. For safety, intraoperative adverse events and 30-day morbidity. For efficacy, successful completion of predefined procedural steps without conversion. The transanal surgical platform consists of a single-port robotic system, while the transabdominal approach can be performed laparoscopically or with single-port robotic assistance.

DETAILED DESCRIPTION:
The study assessed the intraoperative adverse events (device-related and/or procedure-related), postoperative complications, perioperative recovery outcomes, surgical specimen quality, and pathological indices of SPr-taTME in the treatment of mid-to-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Mid or low rectal cancer, 0-10 cm from the anal verge (MRI definition); (2) Histological biopsy showing adenocarcinoma; (3) Stage I-III (MRI and abdominal CT), including the downstaged after neoadjuvant therapy; (4) Intention for primary anastomosis; (5) Obtain the informed consent of the patient and his family; (6) Suitable for robotic or laparoscopic surgery. (7) Over 18 years old.

Exclusion Criteria:

1. T3 tumour with margins less than 1 mm to the mesorectal fascia or T4 tumour, determined by MRI-scan (staged after (chemo)radiotherapy if applicable) ;
2. The anal sphincter complex or levator anal muscle is involved;
3. Previous prostate or rectal surgery (excluding local excision) ;
4. Emergency surgery was performed due to complications of a rectal tumor;
5. Malignancy other than adenocarcinoma at histological examination;
6. Pregnancy;
7. Signs of acute intestinal obstruction;
8. Multiple colorectal tumours;
9. Familial Adenomatosis Polyposis Coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative colitis;
10. Planned synchronous abdominal organ resections;
11. Other malignancies in medical history, except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri;
12. Absolute contraindication to general anaesthesia or prolonged pneumoperitoneum, as severe cardiovascular or respiratory disease (ASA class > III)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative adverse events and 30-day postoperative complications | Intraoperative and postoperative 30 days
  Intraoperative adverse events (device and/or procedure-related). Events were recorded as Preferred Term and classified under System Organ Class as per MedDRA Common Terminology Criteria for Adverse Events (CTCAE) coding guidelines (https://evs.nci.nih.gov/ftp1/CTCAE/About.html). Postoperative complications will refer to any medical occurrence directly attributed to the surgical procedure within the first 30 days.
Conversion rate | Intraoperative
  Conversion to open or laparotomy surgery due to intraoperative complications , technical difficulties, or inability to successfully complete predefined procedural steps .

SECONDARY OUTCOMES:
Quality of specimen (as proposed and published by Quirke et al) | 7 days after surgery
  Quality of specimen (as proposed and published by Quirke et al)
Operative time | Date of surgery (Day 1)
  Record the total operation time, robotic docking time, transanal TME dissection time, and transabdominal TME dissection time respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Li, MD, Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Huichao Zheng, Chongqing, China

IPD SHARING:
Plan to Share IPD: No